CLINICAL TRIAL: NCT04653636
Title: Clinical and MRI Predictive Factors of the Response to Arthrographic Distension and Intensive Physiotherapy in Severe Capsulitis: Improvement of Pain and Function at 1 Month
Brief Title: MRI and Clinical Predictive Factors of the Response to Arthrographic Distension in Severe Capsulitis
Acronym: IRCAP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190073
Record Dates: First submitted 2020-11-19; First posted 2020-12-04 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adhesive capsulitis: Patients presenting to the physical medicine and rehabilitation department [tertiary care] of Cochin Hospital with a clinically diagnosis of severe adhesive capsulitis for whom first-line medical treatment is not effective.
  Interventions: Other: Arthrographic distension; Other: Immediate joint mobilization

INTERVENTIONS:
Other: Arthrographic distension — The treatment consists in one to three shoulder joint capsule arthrographic distension. It consists after local anesthesia, in an injection under pressure of xylocaine 1% and physiological serum in the glenohumeral joint associated with an ampoule of corticosteroids (Betamethasone or Triamcinolone hexacetonide ) at the end of the operation.
  * first arthrographic distension is performed under scopic guidance
  * second and/or third arthrographic distension are performed under ultrasound guidance
  Other Names: Shoulder joint capsule arthrographic distension
Other: Immediate joint mobilization — This procedure was associated with intensive (immediate mobilization, recovery of maximum amplitudes by the physiotherapist and on arthro-motor).
  Physical treatment aimed at rapid amplitude gain and is started immediately after the arthrographic distension, under the effect of local anesthesia. It is at best continued daily at a rate of 2 to 8 hours per day for one to 2 weeks. Depending on the effect obtained on pain and the daily progression of rehabilitation, arthrographic distension may be repeated once or twice during the mobilization period.
  Other Names: Intensive mobilization

SUMMARY:
The purpose of this study is to identify clinical and MRI factors associated to a better response to arthrographic distension in patients with severe capsulitis.

DETAILED DESCRIPTION:
Patients presenting to the physical medicine and rehabilitation department [tertiary care] of Cochin Hospital for severe adhesive capsulitis for whom first-line medical treatment is not effective. The first-line treatment including analgesic, NSAIDs and / or intra-articular infiltration of a corticosteroid derivative and multi-weekly physiotherapy

These patients are integrated into a usual protocol (routine care) consisting of performing an MRI with intravenous injection of gadolinium to confirm the diagnostic and eliminated others causes of shoulder stiffness. IV gadolinium-enhanced MRI can increase the performance of the signal analysis changes of the Synovium and capsule in the Axillary Recess and Rotator interval as compared with unenhanced measures The treatment consists in one to three arthrographic distensions by physiological serum, xylocaine 1% and injection of an ampoule of corticosteroids (DIPROSTENE) associated with intensive (immediate mobilization, recovery of maximum amplitudes by the physiotherapist and on arthro-motor). The primary objective of arthrographic distension is the expansion and rupture of the glenohumeral capsule in the subscapularis recess. It consists after local anesthesia, in an injection under pressure of air or liquid - opacifier or physiological serum - in the glenohumeral joint associated with an infiltration of cortisone derivatives at the end of the operation. Physical treatment aimed at rapid amplitude gain is started immediately after the arthrographic distension, under the effect of local anesthesia. It is at best continued daily at a rate of 2 to 8 hours per day for one to 2 weeks. Depending on the effect obtained on pain and the daily progression of rehabilitation, arthro-distension may be repeated once or twice during the mobilization period.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years,
* Symptomatic shoulder (pain or stiffness) for at least 3 months.
* Patient with failure of treatment including at least NSAIDs, analgesics, +/- intra-articular corticosteroid infiltration and physiotherapy.
* Painful shoulder at inclusion (EN > 5)
* Limitation of passive amplitudes of the glenohumeral joint, of at least 25% of 2 of the 3 mobility sectors (lateral arm elevation, anterior elevation and lateral rotation in the RE1 position), compared to the opposite side
* Absence of glenohumeral arthropathy and abarticular calcification on the standard x-ray of both shoulders.
* Affiliation to a social security
* Information and collection of patient consent

Exclusion Criteria

* Obtain patient consent impossible
* Cognitive disorders considered moderate to severe by the investigator
* Unbalanced diabetes mellitus (glycated hemoglobin> 10%)
* Anticoagulant treatment that cannot be interrupted
* Hemostatic disorders (known history, platelet count <120,000, prothrombin level <75%)
* Allergy to xylocaine, Gadolinium, Diprostene
* Biological inflammatory syndrome
* Pregnant woman (beta human chorionic gonadotropin dosage) or breastfeeding
* Language barrier to the integration of a rehabilitation program or the performance of a reliable assessment.
* People under protective measures
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the physical medicine and rehabilitation department [tertiary care] of Cochin Hospital with a clinically diagnosis of severe adhesive capsulitis for whom first-line medical treatment is not effective.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Physical Impairment: numeric verbal scale of pain | 1 month
  self-evaluated numeric verbal scale of pain, ranging from 0 to 10 (lesser is better)

SECONDARY OUTCOMES:
Physical Impairment: numeric verbal scale of night pain | 1 month
  self-evaluated numeric verbal scale of night pain ranging from 0 to 10 (lesser is better)
Physical Impairment: numeric verbal scale of maximum pain | 1 month
  self-evaluated numeric verbal scale of maximum pain ranging from 0 to 10 (lesser is better)
Disability : numeric verbal scale of disability | 1 month
  self-evaluated numeric verbal scale of disability ranging from 0 to 10 (lesser is better)
Physical Impairment : mobility of shoulder joints | 1 month
  mobility and rotation
Psychological Impairment : Hospital Anxiety and Depression Scale (HADS) | 1 month
  Questionnaire possible presence of anxiety and depressive states It contains two 7-item scales: one for anxiety and one for depression both with a score range of 0-21.
Fear-Avoidance Beliefs Questionnaire (FABQ) | 1 month
  Patient reported questionnaire which specifically focuses on how a patient's fear avoidance beliefs about physical activity and work.
  The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs There are two subscales; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24).
Shoulder Pain and Disability Index (SPADI) | 1 month
  self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. Total score ranging from 0 (best) to 100 (worst).
Disabilities of the Arm, Shoulder and Hand (DASH) | 1 months
  Self-administered questionnaire assessing quality of life of the upper limb. It assesses the ability to perform 23 activities, the severity of symptoms 30-item self-reported questionnaire in which the response options are presented as 5-point Likert scales.
  Scores range from 0 (no disability) to 100 (most severe disability). In addition there are two optional modules of four questions each, sporting or instrumental and employment activity.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Martine LEFEVRE-COLAU, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Rééducation et de Réadaptation de l'Appareil Locomoteur et des Pathologies du Rachis, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No